CLINICAL TRIAL: NCT02658032
Title: Personalized Intervention Program: Tobacco Treatment for Patients at Risk for Lung Cancer (PIP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1505015965; 1P50CA196530-01 (NIH)
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Smoking Cessation; Biofeedback
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard Care/No Bio Feedback (Other): This arm will consist of those first randomized to be enrolled in the standard care arm and then those enrolled in the non bio feedback arm.
  Interventions: Other: standard care
- Standard Care/ Bio Feedback (Other): This arm will consist of those first randomized to be enrolled in the standard care arm and then those enrolled in the bio feedback arm.
  Interventions: Behavioral: bio feedback; Other: standard care
- Personalized Care/ No Bio Feedback (Other): This arm will consist of those first randomized to be enrolled in the personalized care arm and then those enrolled in the non bio feedback arm.
  Interventions: Behavioral: personalized cessation care; Other: standard care
- Personalized Care/ Bio Feedback (Experimental): This arm will consist of those first randomized to be enrolled in the personalized care arm and then those enrolled in the bio feedback arm.
  Interventions: Behavioral: personalized cessation care; Behavioral: bio feedback

INTERVENTIONS:
Behavioral: personalized cessation care — Individuals randomized to this condition will receive standard care (i.e., 5 counseling sessions and nicotine patch(NRT)) and 4 personalized videos with 5 packages of personalized print materials
  Arms: Personalized Care/ Bio Feedback; Personalized Care/ No Bio Feedback
Behavioral: bio feedback — Individuals randomized to this group will be provided with a personalized graph of their biomarker data from baseline, 6 and 8 weeks at the 8-week and 3-month study visits.
  Arms: Personalized Care/ Bio Feedback; Standard Care/ Bio Feedback
Other: standard care
  Arms: Personalized Care/ No Bio Feedback; Standard Care/ Bio Feedback; Standard Care/No Bio Feedback

SUMMARY:
The purpose of this study is to test the efficacy of two separate, sequential interventions to promote tobacco cessation/reduction in patients who are screened for lung cancer or are eligible for lung cancer screening. Each intervention will be compared to standard of care. The first intervention will be a personalized message intervention, the second intervention will consist of a biofeedback-based intervention.

DETAILED DESCRIPTION:
The primary aims of this study are to test the efficacy two types of smoking cessation methods (compared to standard care).

The aim of the first intervention is to evaluate the efficacy of a personalized message intervention in improving tobacco quit rates above and beyond standard care smoking cessation treatment in patients at risk for lung cancer. Messages will be designed specifically for patients at risk for lung cancer, personalized and presented in a gain-framed manner, taking into account demographics and smoking history.

The aim of the second intervention is to evaluate the efficacy of a novel, biofeedback-based intervention that provides personalized individual-level feedback on biomarkers of lung cancer risk and how they improve in response to cessation, delivered in a gain-framed way. The biomarkers include skin carotenoid status, spirometry, and plasma bilirubin, all of which improve with cessation. The study team will examine whether the biofeedback prevents relapse in those who quit and leads to reductions in smoking in lung nodule patients who failed to quit.

Additionally, this study will attempt to evaluate the impact of smoking cessation on miRNA profiles in human serum, especially miRNAs in the let-7 family, which are known to have tumor suppressor function, and which we hypothesize increase in response to cessation.

ELIGIBILITY:
Inclusion Criteria:

* Current Smoker.
* 20 pack per year smoking history.
* Eligible for the Smilow treatment program.
* Willing to enroll in smoking cessation program.
* Willing to be randomized in smoking cessation study.
* English speaking.

Exclusion Criteria:

* Dementia or current serious psychiatric or unstable medical illness.
* Pregnancy or breast feeding.
* Known fat malabsorption diseases that may affect skin carotenoid status.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation | 8 weeks
  Smoking cessation will be measured by self report and validated by the study team using Carbon Monoxide (CO) levels. CO will be measured.
Number of cigarettes smoked | 6 months
  Number of cigarettes smoked will be assessed by self report. Smoking cessation will be measured by self report and validated by the study team using Carbon Monoxide (CO) levels. CO will be measured.

SECONDARY OUTCOMES:
Smoking Cessation | Baseline, 4 Weeks, 3 Months
  Smoking cessation will be measured by self report and validated by the study team using Carbon Monoxide (CO) levels. CO will be measured.
Expired Air | Screening (1 week prior to baseline), Baseline, 8 Weeks, 3 Months, 6 Months
  A hand held spirometer will be used to measure the volume of air expired by the lungs.
Skin Carotenoids | Screening (1 week prior to baseline), Baseline, 6 Weeks, 8 Weeks, 3 Months, 6 Months
  Skin carotenoids are measured with a 30-second scan of the skin with visible light can be used to quantify skin carotenoids rapidly and non-invasively. This study's method sufficiently measures carotenoid status in skin as a biomarker of response to a smoking cessation intervention.
Plasma Bilirubin | Screening (1 week prior to baseline), 6 Weeks, 8 Weeks, 3 Months, 6 Months
  3 mls of blood will be drawn into heparinized tubes, centrifuged, and plasma transferred to opaque tubes and analyzed on the Roche DPP Modular automated chemistry analyzer at the clinical lab, using the method of Jendrassik and Grof. While indirect (unconjugated) bilirubin is likely more relevant for health effects, it is very highly correlated with total bilirubin, which is more common for physicians to test and thus more relevant for translational purposes. Thus, total bilirubin will be used for feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Cartmel, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Medical University of South Carolina: Hollings Cancer Center, Charleston, South Carolina

REFERENCES:
- [Derived] Cartmel B, Fucito LM, Bold KW, Neveu S, Li F, Rojewski AM, Gueorguieva R, O'Malley SS, Herbst RS, Toll BA. Effect of a Personalized Tobacco Treatment Intervention on Smoking Abstinence in Individuals Eligible for Lung Cancer Screening. J Thorac Oncol. 2024 Apr;19(4):643-649. doi: 10.1016/j.jtho.2023.11.012. Epub 2023 Nov 15. PMID 37977486